CLINICAL TRIAL: NCT05627947
Title: Comparison Between Topical Mitomycin C and Cyclosporine After Primary Pterygium Surgery
Brief Title: Comparison Between Topical Mitomycin C and Cyclosporine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMNEYA HEGAZY
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Mitomycin; Cyclosporine

STUDY DESIGN:
Intervention Model Description: compare the recurrence rates and complications associated with instillation of topical mitomycin C and cyclosporine after primary pterygium surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mitomycine-C Group (Active Comparator): This is the First Group and consists of !9 Patients and received 0.02% topical mitomycine C , 4 times per day for five days after the surgery.
  Interventions: Drug: Mitomycin c
- Cyclosporine Group (Active Comparator): This is the Second Group and consists of !9 Patients and received topical 0.05% Cyclosporine, 4 times per day for three months after the surgery.
  Interventions: Drug: Mitomycin c
- artificial eye drops Group (Active Comparator): This is the Third Group and consists of !9 Patients and received artificial eye drops, 4 times per day for three months after the surgery.
  Interventions: Drug: Mitomycin c

INTERVENTIONS:
Drug: Mitomycin c — Comparing the effect of Mitomycin C versus Cyclosporine after primary pterygium surgery
  Other Names: Cyclosporine

SUMMARY:
Pterygium is a disease associated with proliferation of the fibrovascular tissues of the conjunctiva into the cornea and is related to factors such as ultraviolet light exposure, chronic stimulation, inflammation, climate, and genetics.

DETAILED DESCRIPTION:
The first line of treatment for primary pterygium is surgical excision, and despite postoperative adjuvant therapy using mitomycin C, cyclosporine, β-irradiation, argon laser, and bevacizumab, recurrence rates remain high .

Mitomycin C is a metabolic inhibitor extracted from Streptomyces caespitosus that inhibits DNA synthesis .

Cyclosporine is an immunosuppressant that selectively suppresses T-helper cells, controls interleukin synthesis and secretion, and inhibits vascular endothelial growth factor (VEGF)

Bevacizumab is an anti-VEGF antibody that inhibits angiogenesis. Each agent has been studied as an adjuvant therapy to inhibit post-surgery pterygium recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary pterygium
* Pterygium size > or equal 2mm (the horizontal length of the tissue from limbus to cornea will be measured by slit lamp biomicroscopy).
* Ocular discomfort refractory to medical treatment.
* Visual loss induced by pterygium.
* Adult Egyptian population

Exclusion Criteria:

* Patients who had recurrent pterygium or allergy to topical Cyclosporine.
* Patients who had allergy from Mitomycin C.
* Pregnant women.
* Patients with uncontrollable systemic diseases such as hypertension, diabetes, or cardiovascular diseases.
* Patients with diseases of the eye surface such as conjunctivitis and keratitis.
* Patients with a history of eye surgery within the previous six months.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Post Operative recurrence of pterygium | from baseline to 3 months after primary pterygium surgery.
  According to the anterior segment slit lamp examination, grade 0 will be defined as no recurrence; grade 1 will be defined as thin episcleral blood vessels, not accompanied by fibrosis, observed around the excised area; grade 2 will be defined as fibrovascular proliferation limited to the sclera in the area will be excised; grade 3 will be defined as fibrovascular proliferation crossing the corneal limbus. Grades 2 and 3 will be defined as recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Zaki, Assist.Prof., Study Chair — Department of ophthalmology Faculty of Medicine, Menoufia University
Locations (1):
- Faculty of Medicine, Menoufia University, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No